CLINICAL TRIAL: NCT03410927
Title: A Phase 1/2, Open Label, Multicenter Study to Investigate the Safety, Pharmacokinetics, and Efficacy of TAS0728, an Oral Covalent Binding Inhibitor of HER2, in Subjects With Advanced Solid Tumors With HER2 or HER3 Abnormalities
Brief Title: A Study of TAS0728 in Patients With Solid Tumors With HER2 or HER3 Abnormalities
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was stopped due to unacceptable toxicity during the dose-escalation portion (Phase 1) of the study and did not progress to Phase 2
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TO-TAS0728-101; 2017-004415-39 (EudraCT Number)
Record Dates: First submitted 2018-01-19; First posted 2018-01-25 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Advanced Solid Tumors With HER2 Abnormalities; Advanced Solid Tumors With HER3 Abnormalities
Keywords: Phase I; solid tumors; pharmacokinetics; pharmacodynamics; MTD; TAS0728; HER2; HER3 mutation; amplification or overexpression; Urothelial cancer with HER2 or HER3 mutation; Biliary tract cancer with HER2 or HER3 mutation; MBC with HER2 amplification or overexpression or HER3 mutation; NSCLC with HER2 or HER3 mutation; CRC with HER2 or HER3 mutation; amplification
MeSH Terms: interventions — TAS0728

STUDY DESIGN:
Intervention Model Description: In Phase 1, TAS0728 will be evaluated for safety and tolerability, and in phase 2 will be evaluated preliminary efficacy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TAS0728 (Experimental): Group 1: Urothelial cancer with HER2 or HER3 mutation Group 2: Biliary tract cancer with HER2 or HER3 mutation Group 3: Breast cancer with HER2 or HER3 mutation Group 4: Breast cancer with HER2 amplification or overexpression as per American Society of Clinical Oncology - College of American Pathologists (ASCO-CAP) 2013 guidelines Group 5: Non-small cell lung cancer (NSCLC) with HER2 or HER3 mutation Group 6: Colorectal cancer (CRC) with HER2 mutation or amplification Group 7: Other tumors with HER2 or HER3 mutation, amplification, or overexpression (eg, gastric or gastroesophageal junction (GEJ), endometrial)
  Interventions: Drug: TAS0728

INTERVENTIONS:
Drug: TAS0728 — TAS0728 is an oral HER2 covalent inhibitor investigated in patients with advanced solid tumor harboring HER2 or HER3 abnormalities. It will be administered orally at a starting dose of 50 mg BID each morning and evening and escalated to the DLT. The MTD will be used for the phase 2 arms of the study.

SUMMARY:
This is a First-in-Human (FIH), 2-part, Phase 1/2, open-label, multicenter study design to evaluate the safety, tolerability, PK, pharmacodynamics, PGx, and efficacy of TAS0728. This study consists of Phase 1 and Phase 2 components in subjects with advanced solid tumors with HER2 or HER3 overexpression, amplification, or mutation who have progressed despite standard therapy or for which no standard therapy exists, particularly urothelial cancer, biliary tract cancer, metastatic breast cancer, non-small cell lung cancer and colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Male or females with an age ≥ 18 years.
2. Subjects with histological- or cytological-confirmed, advanced cancer, who have progressed on (or not been able to tolerate) standard therapy or for whom no standard anticancer therapy exists

   1. For Phase 1, only subjects HER2 or HER3 molecular/genetic alterations will be enrolled.
   2. For Phase 2a, subjects with one of the following tumor types will be enrolled:

   i. Urothelial cancer with HER2 or HER3 mutation ii. Biliary tract cancer with HER2 or HER3 mutation iii. Breast cancer with HER2 or HER3 mutation iv. Breast cancer with HER2 amplification or overexpression v. NSCLC with HER2 or HER3 mutation vi. CRC with HER2 mutation or amplification vii. Other tumors with HER2 mutation/amplification/overexpression or HER3 mutation (gastric/GEJ, endometrial).
3. At least 1 measurable lesion for solid tumor
4. Is able to take medications orally (e.g., no feeding tube).
5. Able to agree to and sign informed consent and to comply with the protocol
6. Has adequate organ function

Exclusion Criteria:

1. Has a serious illness or medical condition(s)
2. Has received treatment with any proscribed treatments within specified time frames prior to study drug administration
3. Impaired cardiac function or clinically significant cardiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-04-06 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2022-06-09 (Actual)

PRIMARY OUTCOMES:
Number of patients experiencing Dose Limiting Toxicity graded according to CTCAE Version 4.03, observed in the Cycle 1 in order to meet the objective of assessment of the MTD of TAS0728. | 21-day cycles
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] (Phase 1 and 2) | Safety monitoring will begin at the informed consent obtained and continue up to 30 days after the last dose of TAS0728 or until new antitumor therapy, whichever is earlier.
Objective Response Rate using Response Evaluation Criteria in Solid Tumors 1.1 (RECIST) (Phase2) | 3 years

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) after administration of TAS0728 (Phase 1) | 21 days in Cycle 1
Area under the plasma drug concentration-time curve (AUC) after administration of TAS0728 (Phase 1) | 21 days in Cycle 1
Disease Control Rate using RECIST 1.1 (phase 1 and 2) | 3 years
Progression free survival (phase 1 and 2) | 3 years
Duration of response (phase 1 and 2) | 3 years
Overall survival (phase 1 and 2) | 3 years

CONTACTS AND LOCATIONS:
Locations (8):
- United States (5):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Winship Cancer Institute, Atlanta, Georgia
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Sarah Cannon, Nashville, Tennessee
  - University of Texas - MD Anderson, Houston, Texas
- Institut de Cancerologie Gustavo Roussy, Paris, France
- Hospital Vall D'hebron, Barcelona, Spain
- Sarah Cannon Research Institute - UK, London, United Kingdom

REFERENCES:
- [Derived] Piha-Paul SA, Azaro A, Arkenau HT, Oh DY, Galsky MD, Pal SK, Hamada K, He Y, Yamamiya I, Benhadji KA, Hollebecque A. A first-in-human phase I study of TAS0728, an oral covalent binding inhibitor of HER2, in patients with advanced solid tumors with HER2 or HER3 aberrations. Invest New Drugs. 2021 Oct;39(5):1324-1334. doi: 10.1007/s10637-021-01104-7. Epub 2021 Mar 27. PMID 33774767
- [Derived] Irie H, Ito K, Fujioka Y, Oguchi K, Fujioka A, Hashimoto A, Ohsawa H, Tanaka K, Funabashi K, Araki H, Kawai Y, Shimamura T, Wadhwa R, Ohkubo S, Matsuo K. TAS0728, A Covalent-binding, HER2-selective Kinase Inhibitor Shows Potent Antitumor Activity in Preclinical Models. Mol Cancer Ther. 2019 Apr;18(4):733-742. doi: 10.1158/1535-7163.MCT-18-1085. Epub 2019 Feb 20. PMID 30787176